CLINICAL TRIAL: NCT06081296
Title: Dimensional Changes After Different Alveolar Ridge Preservation Techniques for Posterior Region: Randomized Controlled Trial
Brief Title: Dimensional Changes in Alveolar Ridge Preservation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Renato Casarin (Other)
Responsible Party: Sponsor-Investigator, Renato Casarin, Associated Professor, University of Campinas, Brazil
Organization: University of Campinas, Brazil (Other)
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 59208422.8.0000.5418
Record Dates: First submitted 2023-10-02; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization by electronically generated list; Different examiners than operator; Bliding patient;
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Experimental): Alveolus closure with total flap elevation and simple suture
  Interventions: Procedure: Control group
- Group Free Gingival Mixed Graft (Active Comparator): Closure of the alveolus without flap elevation, and placement of a mixed free gingival tissue graft (epithelialized in the central region and de-epithelialized (2 mm) in the vestibulolingual edges
  Interventions: Procedure: Mixed free gingival graft group
- Bone + Mixed Free Gum Graft Group (Active Comparator): Socket closure without flap elevation, placement of lyophilized bone graft and socket sealing with mixed free gingival tissue graft (as previously described)
  Interventions: Procedure: Bone+ mixed free gingival graft group
- Bone + Titanium Seal Group (Active Comparator): Socket closure without flap elevation, placement of lyophilized bone graft, socket sealing by installing a non-absorbable titanium membrane.
  Interventions: Procedure: Bone + Titanium Seal group

INTERVENTIONS:
Procedure: Control group — Control Group (Ctl): alveolus closure with total flap elevation and simple suture; and socket sealing with mixed free gingival tissue graft.
  Other Names: Mixed free gingival graft group; Bone+ mixed free gingival graft group; Bone + Titanium Seal group
  Arms: Control group
Procedure: Mixed free gingival graft group — closure of the alveolus without flap elevation, and placement of a free gingival tissue graft removed from the individual's own palate, which will be properly sutured. This graft is a combination of epithelialized-subepithelial connective tissue graft, which will be taken from the hard palate of the regions.
  Other Names: Bone+ mixed free gingival graft group; Bone + Titanium Seal group
  Arms: Group Free Gingival Mixed Graft
Procedure: Bone+ mixed free gingival graft group — closure of the socket without flap elevation, placement of a freeze-dried bone graft and sealing of the socket with a mixed free gingival tissue graft.
  Other Names: Bone + Titanium Seal group
  Arms: Bone + Mixed Free Gum Graft Group
Procedure: Bone + Titanium Seal group — socket closure without flap elevation, placement of lyophilized bone graft, socket sealing by installing a non-absorbable titanium membrane.
  Arms: Bone + Titanium Seal Group

SUMMARY:
Objective: The objective is to evaluate the dimensional changes of soft tissue and alveolar ridge after extraction of posterior elements with different clinical protocols of alveolar preservation.

DETAILED DESCRIPTION:
Detailed methodology: 80 individuals will be selected with need for extraction of premolar and molar elements, from both arches, for non-periodontal reasons, to participate in this randomized controlled clinical study. The dental elements will be extracted atraumatically, and allocated to one of the study groups (n=20/grp): Control Group (Ctl): alveolus closure with total flap elevation and simple suture; Group Free Gingival Mixed Graft (EGLM): closure of the alveolus without flap elevation, and placement of a mixed free gingival tissue graft (epithelialized in the central region and de-epithelialized (2 mm) in the vestibulolingual edges;

Bone + Mixed Free Gum Graft Group (B+EGLM): socket closure without flap elevation, placement of lyophilized bone graft and socket sealing with mixed free gingival tissue graft (as previously described);

Bone + Titanium Seal Group (B+TS): socket closure without flap elevation, placement of lyophilized bone graft, socket sealing by installing a non-absorbable titanium membrane. Immediately after the extractions, Cone Beam Computed Tomography (90 kVp/8 mA/2.3 sec) will be performed, with lip/cheek separation, with 1.5 mm thick slices and a 1 mm distance, with a field of vision (FOV) of 5±5 cm, which will be repeated after 6 months. During the CT scans, the patients will use intra-oral appliances with hyperdense indicators to determine the reference points to measure the variables: bone tissue height in the center of the socket (primary variable) and every 2 mm equidistantly; thickness of bone tissue in the center of the socket and every 2 mm equidistantly. Soft tissue variables will also be evaluated, such as: mucosal thickness at the height and 2 mm below the edge margin (by CT); height of the keratinized tissue (measured by a dry tip caliper). After 6 months, all patients will receive dental implants, with the ideal measurements for bone dimension, and the possibility of installing implants >10mm or <10mm in length will be statistically analyzed. After 4 months of dental implant placement, single prostheses will be installed and CT, soft tissue measurements and clinical parameters will be repeated (peri-implant depth; presence of biofilm and bleeding on probing; tissue thickness at the margin and 2 mm below; keratinized tissue). Implants will be re-evaluated after 12 months. All measurements will be performed by a previously calibrated examiner (intra-class correlation above 90%). The data will initially be analyzed in a descriptive way, with means and standard deviations. For comparison between groups and times, two-way/Tukey ANOVA test will be used. In all analyses, a significance level of 5% will be considered.

ELIGIBILITY:
Inclusion Criteria:

* Systemic health (Hypertension and Diabetes controlled)
* Indication of tooth extraction with at least 2/3 of the bone support, in the premolar or molar region
* Signing the consent form
* Individuals over 18 years of age.

Exclusion Criteria:

* Presence of periodontal disease at the time of surgery
* Pregnant and lactating women
* Smokers
* Being in orthodontic treatment
* Use medication that alters the bone healing process, such as those used to treat osteoporosis and the bisphosphonate group
* Individuals under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-10-15 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
assessment of dimensional change using linear measurements through CT, evaluating bone remodeling. | 6 months
  Through CT taken immediately after tooth extraction and six months later, these images will be analyzed to evaluate changes in hard tissues

SECONDARY OUTCOMES:
evaluation of the dimensional change of soft tissues that accompany bone remodeling through linear and volume measurements in the STL | 6 months
  Through STLs taken immediately after extraction and six months later, these images will be analyzed to evaluate changes in soft tissues
Visual analogy scale for pain and disconfort evaluattion which consists of a score to measure the patient's pain intensity. | 1 week
  Will be also evaluate post-operative pain and discomfort,.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Casarin, PhD, Principal Investigator — University of Campinas, Brazil
Locations (1):
- Piracicaba Dental School, Piracicaba, São Paulo, Brazil

REFERENCES:
- [Derived] Sandoli Arroteia L, Lopes MP, Rea MT, Vieira E Oliveira TR, Oliveira ML, de Faveri M, Santamaria MP, Queiroz LA, Casati MZ, Casarin RCV. Dimensional Changes After Different Alveolar Ridge Preservation Techniques for Posterior Region: A Randomised Controlled Clinical Trial. J Clin Periodontol. 2025 Nov;52(11):1584-1594. doi: 10.1111/jcpe.70004. Epub 2025 Aug 5. PMID 40762250